CLINICAL TRIAL: NCT03577834
Title: The Effect of Vinegar Consumption on Visceral Fat and Blood Glucose Concentration
Acronym: VIVO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carol Johnston (Other)
Responsible Party: Sponsor-Investigator, Carol Johnston, Professor and Associated Director, Arizona State University
Organization: Arizona State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: vinegar_visceral_fat
Record Dates: First submitted 2018-06-25; First posted 2018-07-05 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Visceral Obesity; Tooth Erosion; Insulin Resistance
Keywords: randomized clinical trial; vinegar; adiposity; insulin resistance
MeSH Terms: conditions — Obesity, Abdominal; Tooth Erosion; Insulin Resistance; Obesity | interventions — Acetic Acid

STUDY DESIGN:
Intervention Model Description: Qualifying participants will be stratified by gender, age, weight, and waist circumference, then randomized into two groups: the intervention group, vinegar drinks (VIN) or the control group, vinegar pills (CON).
Who Masked: Participant, Investigator
Masking Description: All participants will receive 'vinegar' either in liquid form (active) or pill (not active as acetic acid concentration is below threshold of effect). Investigators measuring outcome variables (visceral fat, tooth enamel, and blood indices) are blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liquid vinegar (Experimental): Participants in this arm were instructed to drink 2 tablespoons of red wine vinegar (provided) mixed with water twice each day for weeks 1 to 8 of the trial.
  Interventions: Dietary Supplement: liquid vinegar
- Vinegar pill (Placebo Comparator): Participants in the control group were instructed to take one vinegar pill (provided) each day for weeks 1-8 of the trial.
  Interventions: Dietary Supplement: vinegar pill

INTERVENTIONS:
Dietary Supplement: liquid vinegar — 6% red wine vinegar (2 tablespoons providing 1.7 g acetic acid)
  Other Names: VIN
  Arms: Liquid vinegar
Dietary Supplement: vinegar pill — Apple Cider Vinegar Tablets (1 tablet providing 0.0225 g acetic acid)
  Other Names: CON
  Arms: Vinegar pill

SUMMARY:
The purpose of this study is to test the potential ability of vinegar to significantly decrease visceral fat in healthy adults with "central obesity". During the 8-week trial, participants will either consume a low-dose vinegar pill (control treatment) or a vinegar drink twice per day.

Research Aim and Hypothesis H1 Daily vinegar consumption will be associated with loss in visceral fat (as measured by DXA) after 8 weeks compared to the placebo treatment (low-vinegar pill) in a group of healthy adults with "central obesity".

H2 Daily vinegar consumption will be associated with a decrease in abdominal circumference after 8 weeks compared to the placebo treatment (low-vinegar pill) in a group of healthy adults with "central obesity".

DETAILED DESCRIPTION:
This randomized, placebo-controlled experimental trial will last 8 weeks. At the initial visit (consenting visit lasting about 20 minutes) the participant will sign the consent and complete a short health questionnaire and a short questionnaire on tooth erosion. Body height and weight and waist circumference will also be measured. Qualifying participants will be stratified by gender, age, weight, and waist circumference, then randomized into two groups: the intervention group, vinegar drinks (VIN) or the control group, vinegar pills (CON). The participants will know which treatment they are given but they will not know which group (control vs. placebo) they are in. Those who receive the VIN will be instructed to drink 2 tablespoons of red wine vinegar (provided) mixed with water twice each day for weeks 1 to 8 of the trial. Those in the CON group will be instructed to take one vinegar pill (provided) each day for weeks 1-8 of the trial. Participants will be instructed to maintain their current diet and exercise habits during the study.

ELIGIBILITY:
Inclusion Criteria:

* Nonsmoking
* Not pregnant or lactating if female
* No active disease state or medication use affecting blood glucose or cholesterol (additionally, individuals on digoxin or diuretics will be excluded but other medications in use >3 months will be allowed)
* No food restrictions or special diet
* BMI range: 22-35
* Waist circumference >34 (women) and >39 (males)
* Sedentary (exercising < 3 days/week)

Exclusion Criteria:

* Unwilling to take a vinegar supplement daily for 8 week or follow other aspects of study protocol
* Recent abdominal surgery or condition causing abdominal discomfort/distention (such as acid reflux, ascites, pancreatitis, diverticulitis/diverticulosis, Crohn's disease, and/or irritable bowel syndrome)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
visceral adiposity | change after 8 weeks of treatment
  visceral fat as measured by DXA

SECONDARY OUTCOMES:
tooth erosion | change after 8 weeks of treatment
  dental exam using Basic Erosion Wear Examination (BEWE)
insulin resistance | change after 8 weeks of treatment
  measurement of insulin resistance using HOMA-IR (fasting glucose and fasting insulin index)

REFERENCES:
- [Derived] Anderson S, Gonzalez LA, Jasbi P, Johnston CS. Evidence That Daily Vinegar Ingestion May Contribute to Erosive Tooth Wear in Adults. J Med Food. 2021 Aug;24(8):894-896. doi: 10.1089/jmf.2020.0108. Epub 2020 Dec 9. PMID 33297831